CLINICAL TRIAL: NCT00588770
Title: A Phase III Randomized Trial of Chemotherapy With or Without Bevacizumab in Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: Chemotherapy With or Without Bevacizumab in Treating Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00507; NCI-2009-00507 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1305; CDR0000582533; E1305 (Other: ECOG-ACRIN Cancer Research Group); E1305 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-09 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Neck Squamous Cell Carcinoma of Unknown Primary; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Neck Squamous Cell Carcinoma of Unknown Primary; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Salivary Gland Carcinoma; Recurrent Sinonasal Squamous Cell Carcinoma; Salivary Gland Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Major Salivary Gland Cancer AJCC v7; Stage IVA Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Laryngeal Verrucous Carcinoma AJCC v7; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Major Salivary Gland Cancer AJCC v7; Stage IVA Oral Cavity Cancer AJCC v6 and v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Sinonasal Squamous Cell Carcinoma AJCC v7; Stage IVB Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Laryngeal Verrucous Carcinoma AJCC v7; Stage IVB Lip and Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVB Major Salivary Gland Cancer AJCC v7; Stage IVB Oral Cavity Cancer AJCC v6 and v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Sinonasal Squamous Cell Carcinoma AJCC v7; Stage IVC Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Laryngeal Verrucous Carcinoma AJCC v7; Stage IVC Lip and Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVC Major Salivary Gland Cancer AJCC v7; Stage IVC Oral Cavity Cancer AJCC v6 and v7; Stage IVC Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Sinonasal Squamous Cell Carcinoma AJCC v7; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Fluorouracil; dehydroftorafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Arm IA (docetaxel, cisplatin) (Active Comparator): Patients receive docetaxel IV over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm IB (docetaxel, cisplatin, bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and docetaxel and cisplatin as in Arm IA.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm IIA (docetaxel, carboplatin) (Active Comparator): Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm IIB (docetaxel, carboplatin, bevacizumab) (Experimental): Patients receive bevacizumab as in Arm IB and docetaxel and carboplatin as in Arm IIA.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis
- Arm IIIA (cisplatin, fluorouracil) (Active Comparator): Patients receive cisplatin IV over 1-2 hours on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis
- Arm IIIB (cisplatin, fluorouracil, bevacizumab) (Experimental): Patients receive bevacizumab as in Arm IB and cisplatin and fluorouracil as in Arm IIIA.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis
- Arm IVA (carboplatin, fluorouracil) (Active Comparator): Patients receive carboplatin IV over 30 minutes on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis
- Arm IVB (carboplatin, fluorouracil, bevacizumab) (Experimental): Patients receive bevacizumab as in Arm IB and carboplatin and fluorouracil as in Arm IVA.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm IB (docetaxel, cisplatin, bevacizumab); Arm IIB (docetaxel, carboplatin, bevacizumab); Arm IIIB (cisplatin, fluorouracil, bevacizumab); Arm IVB (carboplatin, fluorouracil, bevacizumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm IIA (docetaxel, carboplatin); Arm IIB (docetaxel, carboplatin, bevacizumab); Arm IVA (carboplatin, fluorouracil); Arm IVB (carboplatin, fluorouracil, bevacizumab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm IA (docetaxel, cisplatin); Arm IB (docetaxel, cisplatin, bevacizumab); Arm IIIA (cisplatin, fluorouracil); Arm IIIB (cisplatin, fluorouracil, bevacizumab)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm IA (docetaxel, cisplatin); Arm IB (docetaxel, cisplatin, bevacizumab); Arm IIA (docetaxel, carboplatin); Arm IIB (docetaxel, carboplatin, bevacizumab)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm IIIA (cisplatin, fluorouracil); Arm IIIB (cisplatin, fluorouracil, bevacizumab); Arm IVA (carboplatin, fluorouracil); Arm IVB (carboplatin, fluorouracil, bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies chemotherapy to see how well it works with or without bevacizumab in treating patients with head and neck squamous cell carcinoma that has come back (recurrent) or that has spread to other parts of the body (metastatic). Drugs used in chemotherapy, such as docetaxel, cisplatin, carboplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab may also make tumor cells more sensitive to chemotherapy and stop the growth of head and neck cancer by blocking blood flow to the tumor. It is not yet known whether combination chemotherapy is more effective when given with or without bevacizumab in treating patients with head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival of patients with recurrent or metastatic head and neck cancer treated with standard platinum-based chemotherapy with or without bevacizumab.

SECONDARY OBJECTIVES:

I. To assess toxicities with the addition of bevacizumab to each platinum-doublet (cisplatin/docetaxel, carboplatin/docetaxel, cisplatin/fluorouracil [5-FU], carboplatin/5-FU).

II. To compare the objective response rates and the progression-free survival achieved with the above therapies.

III. To collect blood samples before and after therapy for future correlative studies.

IV. To collect tumor tissue samples available at baseline from prior diagnostic procedures for future correlative studies.

OUTLINE: After the physician decides which chemotherapy doublet to use, patients are randomized to 1 of 2 treatment arms for that chemotherapy combination.

ARM IA: Patients receive chemotherapy comprising docetaxel intravenously (IV) over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM IB: Patients receive bevacizumab IV over 30-90 minutes on day 1 and docetaxel and cisplatin as in Arm IA.

ARM IIA: Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM IIB: Patients receive bevacizumab as in arm IB and docetaxel and carboplatin as in Arm IIA.

ARM IIIA: Patients receive cisplatin IV over 1-2 hours on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM IIIB: Patients receive bevacizumab as in Arm IB and cisplatin and fluorouracil as in Arm IIIA.

ARM IVA: Patients receive carboplatin IV over 30 minutes on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM IVB: Patients receive bevacizumab as in Arm IB and carboplatin and fluorouracil as in Arm IVA.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell cancer of the head and neck (SCCHN), from any primary site, including unknown primary cancers of the head and neck; patient must not have nasopharyngeal carcinoma of histologic types World Health Organization (WHO) 2 or 3 or squamous cell carcinoma that originated in the skin
* Patients must have SCCHN that is either (a) recurrent, judged incurable by surgery or radiation or (b) metastatic; NOTE: Patients who refuse radical resection for recurrent disease are eligible; NOTE: A second primary squamous cell carcinoma of the head and neck is allowed if eligibility is based on a recurrent or metastatic first primary squamous cell carcinoma of the head and neck
* No prior chemotherapy or biologic/molecular targeted therapy for recurrent or metastatic SCCHN

  * Patients may have received one regimen of induction, concomitant chemoradiotherapy and/or adjuvant chemotherapy as part of initial potential curative therapy but must not have received prior chemotherapy for recurrent or metastatic disease
  * A minimum of 4 months is required between last dose of chemotherapy or chemoradiotherapy and study treatment; in addition patients must be progression-free for at least 4 months after completion of chemotherapy or chemoradiotherapy or radiation plus cetuximab given with a curative intent; (cetuximab therapy: 4 months is required between last dose of chemotherapy or chemoradiotherapy and study treatment if part of concurrent regimen, 8 weeks if part of adjuvant regimen post radiation)
  * Patients having progression after 2 cycles of induction chemotherapy are not eligible for the study
* No prior bevacizumab is allowed
* A maximum of one prior radiotherapy regimen, curative or palliative, to the head and neck is allowed; if the radiation is combined with chemotherapy and/or cetuximab, a minimum of 4 months must elapse between the end of radiotherapy and registration; if the radiation is given alone, a minimum of 8 weeks must elapse between the end of radiotherapy and registration; a minimum of 3 weeks must elapse between prior radiation to other areas and registration
* Patients must not be receiving any other investigational agent while on the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have recovered to grade 1 or better from any acute effects of prior surgery, chemotherapy, or radiation therapy, and should be > 4 weeks post surgery; chronic late xerostomia, speech and swallowing abnormalities resulting from prior radiation or surgery are permitted if nutritional status is stable
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST); baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to randomization; disease in previously irradiated sites is considered measurable if there has been unequivocal disease progression or biopsy-proven residual carcinoma following radiation therapy; persistent disease after radiotherapy must be biopsy proven at least 8 weeks after completion of radiation therapy; (radiographic findings are acceptable providing that clear-cut measurements can be made)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Hemoglobin (Hgb) >= 8.0 g/dL
* Platelet count >= 100,000/mm^3
* Creatinine clearance of >= 60 ml/min; creatinine clearance may be measured or calculated; if calculating, creatinine clearance, use the Cockroft-Gault formula
* Total bilirubin within normal limits (must be obtained =< 2 weeks prior to randomization)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) must be within the range allowing for eligibility

  * Alkaline phosphatase normal AND AST or ALT =< 5 x upper limit of normal (ULN)
  * Alkaline phosphatase > 1 but =< 2.5 x ULN AND AST or ALT > 1 but =< 1.5 x ULN
  * Alkaline phosphatase > 2.5 but =< 5 x ULN AND AST or ALT normal
* Alkaline phosphatase must be within the range allowing for eligibility
* Urine dipstick must be =< 0-1+ within 2 weeks (14 days) of randomization; if urine dipstick result is > 1+, a calculation of urine protein creatinine (UPC) ratio is required; patients must have a UPC ratio < 1.0 to participate in the study; NOTE: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* No known brain metastases
* Patients who meet the following criteria will be excluded:

  * Tumors that invade major vessels (e.g. the carotid) as shown unequivocally by imaging studies
  * Central (i.e. within 2 cm from the hilum) lung metastases that are cavitary as shown unequivocally by imaging studies
  * Any prior history of bleeding related to the current head and neck cancer
  * History of gross hemoptysis (bright red blood of 1/2 teaspoon or more per episode of coughing) =< 3 months prior to enrollment
* No history of coagulopathy or hemorrhagic disorders
* Patients should not have a history of thrombosis (e.g. pulmonary embolism or deep venous thrombosis) currently requiring therapeutic anticoagulation (prophylactic use of warfarin 1 mg per day is allowed) and international normalized ratio (INR) should be < 1.5 at registration
* Patients must not be receiving chronic daily treatment with aspirin (> 325 mg/day) or non-steroidal anti-inflammatory agents (NSAID's) known to inhibit platelet function; the use of anti-platelet agents (e.g. dipyridamole [Persantine], ticlopidine [Ticlid], clopidogrel [Plavix]) is allowed only if patient is not receiving aspirin or NSAID's known to inhibit platelet function
* No hypercalcemia related to head and neck cancer
* Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated; patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post diagnosis
* No current peripheral neuropathy >= grade 2 at time of randomization
* Patients must not have any co-existing condition that would preclude full compliance with the study
* No prior history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80, if the physician's choice of chemotherapy regimen is docetaxel
* All patients must have blood pressure =< 150/90 =< 2 weeks prior to randomization; patients with history of hypertension must be well-controlled upon study entry (=< 150/90) on a stable regimen of anti-hypertensive therapy
* No major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study
* No unstable angina or myocardial infarction within the previous 6 months; no symptomatic congestive heart failure, New York Heart Association (NYHA) grade II or greater; no history of aortic dissection or presence of aneurysm > 6 cm (or at high risk for rupture); no serious cardiac arrhythmia requiring medication (history of chronic atrial fibrillation or other atrial arrhythmia with controlled rate on medication is allowed); no clinically significant peripheral vascular disease manifested by intermittent claudication or need for vascular intervention; no history of aortic dissection; no history of any central nervous system (CNS) cerebrovascular ischemia or stroke within the last 6 months; no active serious infection
* Patients should not have prior history of a serious human anti-human antibody (HAHA) reaction; patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies are not eligible
* Women must not be pregnant or breast feeding; pregnant women are excluded from this study; women of child-bearing potential and men must agree to total abstinence or to use adequate hormonal or barrier method of birth control prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2008-08-08 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios (Ethan) Argiris, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (782):
- United States (780):
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Saint Helena Hospital, St. Helena, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Space Coast Cancer Centers-Titusville, Titusville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Garnet Health Medical Center, Middletown, New York
  - Mount Sinai Union Square, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Southlake Clinic, Renton, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Derived] Argiris A, Li S, Savvides P, Ohr JP, Gilbert J, Levine MA, Chakravarti A, Haigentz M Jr, Saba NF, Ikpeazu CV, Schneider CJ, Pinto HA, Forastiere AA, Burtness B. Phase III Randomized Trial of Chemotherapy With or Without Bevacizumab in Patients With Recurrent or Metastatic Head and Neck Cancer. J Clin Oncol. 2019 Dec 1;37(34):3266-3274. doi: 10.1200/JCO.19.00555. Epub 2019 Oct 16. PMID 31618129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E1305 was activated on August 8, 2008 and closed on February 11,2015, with final accrual of 403 patients.
Groups:
- Chemotherapy Arm (Arm A): ARM A: Patients receive one of the four chemotherapy regimens
  ARM IA: Patients receive chemotherapy comprising docetaxel intravenously (IV) over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IIA: Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IIIA: Patients receive cisplatin IV over 1-2 hours on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IVA: Patients receive carboplatin IV over 30 minutes on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Chemotherapy+Bevacizumab (Arm B): ARM B: Patients receive bevacizumab in addition to the chemotherapy regimen as in arm A
  ARM IB: Patients receive bevacizumab IV over 30-90 minutes on day 1 and docetaxel and cisplatin as in Arm IA.
  ARM IIB: Patients receive bevacizumab as in arm IB and docetaxel and carboplatin as in Arm IIA.
  ARM IIIB: Patients receive bevacizumab as in Arm IB and cisplatin and fluorouracil as in Arm IIIA.
  ARM IVB: Patients receive bevacizumab as in Arm IB and carboplatin and fluorouracil as in Arm IVA.
Period: Overall Study
Arm/Group | Chemotherapy Arm (Arm A) | Chemotherapy+Bevacizumab (Arm B)
Started | 200 | 203
Eligible | 188 | 183
Start Protocol Therapy | 200 | 194
Completed | 41 | 3
Not Completed | 159 | 200
Not completed — Disease progression | 85 | 68
Not completed — Adverse Event | 29 | 58
Not completed — Death | 13 | 22
Not completed — Withdrawal by Subject | 15 | 25
Not completed — Alternative therapy | 2 | 4
Not completed — Other complicating disease | 3 | 2
Not completed — Not start protocol therapy | 0 | 9
Not completed — Lack of Efficacy | 8 | 10
Not completed — Physician discretion | 2 | 0
Not completed — Patient non-compliance | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Arm (Arm A) | Chemotherapy+Bevacizumab (Arm B) | Total
Number analyzed (Participants) | 200 | 203 | 403
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 86] | 58 [29 to 82] | 58 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 168 | 176 | 344
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 168 | 179 | 347
  Black | 21 | 18 | 39
  Other | 4 | 2 | 6
  Not reported | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as time from randomization to death from any course. Patients who were alive were censored at the last contact date. Median OS was estimated using the Kaplan-Meier method.
Time Frame: assessed every 3 months within 2 years from study entry, then every 6 months up to 5 years from study entry
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Chemotherapy+Bevacizumab (Arm B): ARM B: Patients receive bevacizumab in addition to the chemotherapy regimen as in arm A
  ARM IB: Patients receive bevacizumab IV over 30-90 minutes on day 1 and docetaxel and cisplatin as in Arm IA.
  ARM IIB: Patients receive bevacizumab as in arm IB and docetaxel and carboplatin as in Arm IIA.
  Regimen 2:
  ARM IIIB: Patients receive bevacizumab as in Arm IB and cisplatin and fluorouracil as in Arm IIIA.
  Regimen 2 carbo:
  ARM IVB: Patients receive bevacizumab as in Arm IB and carboplatin and fluorouracil as in Arm IVA.
Arm/Group | Chemotherapy Arm (Arm A) | Chemotherapy+Bevacizumab (Arm B)
Number analyzed (Participants) | 200 | 203
months | 11.0 [9.5 to 13.0] | 12.6 [10.3 to 15.8]
Statistical Analysis 1: Comparison: Chemotherapy Arm (Arm A) vs Chemotherapy+Bevacizumab (Arm B); The study hypothesis is that the addition of bevacizumab will improve the median survival by 35% from 8.5 months (based on E1395 and E5397) to 11.5 months; Test type: Superiority; p = 0.22, Log Rank — The P value was based on stratified log rank test, stratified by choice of chemotherapy combination, performance status, weight loss in the last 6 months, and prior radiation of the head and neck

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Progression-free survival (PFS) was defined as the time from randomization to date of disease progression or death from any cause, whichever occurred first. Patients who were still alive and progression free were censored at last disease assessment date. Median PFS was estimated using Kaplan-Meier method.
Time Frame: on both arms, assessed every 2 cycles during chemotherapy treatment, then assessed every 9 weeks until progression up to 5 years from study entry; patients on arm B were assessed every 2 cycles for additional 12 weeks before changing to every 9 weeks
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Arm (Arm A) | Chemotherapy+Bevacizumab (Arm B)
Number analyzed (Participants) | 200 | 203
months | 4.3 [3.8 to 5.2] | 6.0 [4.9 to 6.7]

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by all patients. Responses are evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR is defined as disappearance of all target and non-target lesions. PR is defined as disappearance of target lesions or at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and persistence of one or more non-target lesion(s).
Time Frame: as for outcome 2
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Chemotherapy Arm (Arm A) | Chemotherapy+Bevacizumab (Arm B)
Number analyzed (Participants) | 200 | 203
proportion of participants | 0.245 [0.187 to 0.311] | 0.355 [0.289 to 0.425]

4. Other Pre Specified Outcome: To Collect Blood Samples Before and After Therapy for Future Correlative Studies
Description: These were blood and tissue samples collections and have no data to report.
Time Frame: Before and after therapy
Reporting Status: Not Posted

5. Other Pre Specified Outcome: To Collect Tumor Tissue Samples Available at Baseline From Prior Diagnostic Procedures for Future Correlative Studies
Description: These were blood and tissue samples collections and have no data to report.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed at the end of each cycle (1 cycle=21 days) while on treatment and at 3 months post treatment (to report late adverse events)
Description: At Risk for All-Cause Mortality includes all enrolled participants; at Risk for all other Adverse Events includes the safety population.
  A total of four chemotherapy regimen choices were allowed for the platinum-doublet treatment, and chemotherapy regimen choice was at the discretion of the treating physician and was made prior to randomization. The trial did not intent to look at the four chemotherapy regimens separately in terms of safety and efficacy.
Groups:
- Chemotherapy (Arm A): ARM A: Patients receive one of the four chemotherapy regimens
  ARM IA: Patients receive chemotherapy comprising docetaxel intravenously (IV) over 1 hour and cisplatin IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IIA: Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IIIA: Patients receive cisplatin IV over 1-2 hours on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ARM IVA: Patients receive carboplatin IV over 30 minutes on day 1 and fluorouracil IV continuously on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Chemotherapy + Bevacizumab (Arm B): ARM B: Patients receive bevacizumab in addition to the chemotherapy regimen as in arm A
  ARM IB: Patients receive bevacizumab IV over 30-90 minutes on day 1 and docetaxel and cisplatin as in Arm IA.
  ARM IIB: Patients receive bevacizumab as in arm IB and docetaxel and carboplatin as in Arm IIA.
  ARM IIIB: Patients receive bevacizumab as in Arm IB and cisplatin and fluorouracil as in Arm IIIA.
  ARM IVB: Patients receive bevacizumab as in Arm IB and carboplatin and fluorouracil as in Arm IVA.
Arm/Group | Chemotherapy (Arm A) | Chemotherapy + Bevacizumab (Arm B)
All-Cause Mortality (participants affected / at risk) | 182/200 | 175/203
Serious Adverse Events (participants affected / at risk) | 135/199 | 162/193
Other Adverse Events (participants affected / at risk) | 50/199 | 50/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (Arm A) (N=199) | Chemotherapy + Bevacizumab (Arm B) (N=193)
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 17 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 35
Asystole (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 1 | 2
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 1
Fatigue (General disorders) | 20 | 34
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 7
Colitis (Gastrointestinal disorders) | 0 | 2
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 9
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 9
Esophageal fistula (Gastrointestinal disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 3
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 8 | 37
Nausea (Gastrointestinal disorders) | 15 | 22
Oral hemorrhage (Gastrointestinal disorders) | 0 | 4
Oral pain (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 14
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Cranial nerve infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gum infection (Infections and infestations) | 0 | 2
Kidney infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 5
Mucosal infection (Infections and infestations) | 1 | 0
Salivary gland infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Skin infection (Infections and infestations) | 2 | 3
Soft tissue infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 2
Infections and infestations - Other (Infections and infestations) | 3 | 6
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 1 | 2
Lymphocyte count decreased (Investigations) | 12 | 12
Neutrophil count decreased (Investigations) | 53 | 73
Platelet count decreased (Investigations) | 13 | 15
Weight loss (Investigations) | 4 | 5
White blood cell decreased (Investigations) | 33 | 51
Investigations - Other, specify (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 13 | 12
Dehydration (Metabolism and nutrition disorders) | 11 | 30
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 8 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 6
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Reversible posterior leukoencephalopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 5
Nervous system disorders - Other (Nervous system disorders) | 0 | 2
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 3
Proteinuria (Renal and urinary disorders) | 0 | 3
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 12
Hypotension (Vascular disorders) | 3 | 4
Thromboembolic event (Vascular disorders) | 1 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (Arm A) (N=199) | Chemotherapy + Bevacizumab (Arm B) (N=193)
Fatigue (General disorders) | 13 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 11
Platelet count decreased (Investigations) | 9 | 10
Anorexia (Metabolism and nutrition disorders) | 6 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 28 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT00588770/Prot_SAP_000.pdf